CLINICAL TRIAL: NCT02462200
Title: Shave Margins in Breast Conservation Therapy (SMART): A Randomized Controlled Trial
Brief Title: Shave Margins in Breast Conservation Therapy
Acronym: SMART
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient funding
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201506053
Record Dates: First submitted 2015-06-01; First posted 2015-06-03 (Estimated); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Breast Cancer; Cancer of Breast; Cancer of the Breast
MeSH Terms: conditions — Breast Neoplasms | interventions — Mastectomy, Segmental; Indocyanine Green

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BCS Arm (breast-conserving surgery - standard of care) (Active Comparator): * Defined as partial mastectomy, lumpectomy, or local excisional biopsy with or without needle/wire localization
  * The ICG will be prepared per manufacturer instructions and diluted to allow for intravenous dosing up to 0.5 mg/kg (except for those patients with iodine or seafood allergies or in cases where the goggles are unavailable for use).
  * Following the BCS procedures, the surgeon or a study team member will don the goggles and state the NIR fluorescence margin information of the excised primary tumor specimen and of and CSM that are taken.
  Interventions: Procedure: Breast-conserving surgery (BCS); Behavioral: BREAST-Q Questionnaire; Device: 3-D breast imaging; Other: Indocyanine green; Device: Intraoperative imaging device; Procedure: Peripheral blood draw
- CSM Arm (breast-conserving surgery with cavity shave margins) (Experimental): * Partial mastectomy, lumpectomy, or local excisional biopsy with or without needle/wire localization with the addition of additional tissue specimens from all 6 margins (anterior, posterior, superior, inferior, medial, lateral) of the wound cavity if possible. In cases where an additional margin would involve the skin at the anterior margin and/or the pectoral muscle at the posterior margin, only the 4 (or 5) remaining margins should be obtained
  * A margin thickness of 1 cm will be the defined goal to establish uniformity among different surgeons and allow for appropriate pathological evaluation
  * The ICG will be prepared per manufacturer instructions and diluted to allow for intravenous dosing up to 0.5 mg/kg (no iodine or seafood allergies).
  * Following the BCS procedures, the surgeon or a study team member will don the goggles and state the NIR fluorescence margin information of the excised primary tumor specimen and of any CSM that are taken.
  Interventions: Procedure: Breast-conserving surgery (BCS); Procedure: Cavity shave margins (CSM); Behavioral: BREAST-Q Questionnaire; Device: 3-D breast imaging; Other: Indocyanine green; Device: Intraoperative imaging device; Procedure: Peripheral blood draw

INTERVENTIONS:
Procedure: Breast-conserving surgery (BCS)
Procedure: Cavity shave margins (CSM)
  Arms: CSM Arm (breast-conserving surgery with cavity shave margins)
Behavioral: BREAST-Q Questionnaire
Device: 3-D breast imaging — Using a 3-D breast imaging camera Vectra 3-D XT
Other: Indocyanine green
  Other Names: ICG
Device: Intraoperative imaging device — The goggle device is wearable, compact, and battery-operated, and it allows for hands-free operation by the wearer. The goggles provide functional information via a NIR light-emitting diode (LED) integrated within one of the eyepieces, which causes NIR fluorescence excitation of the molecular probes within the surgical field
Procedure: Peripheral blood draw — -Time of surgery if coordinator is available

SUMMARY:
The investigators propose a randomized controlled superiority trial of standard breast-conserving surgery (BCS) versus BCS with cavity shave margins (CSM). The main objectives of this trial will be to evaluate prospectively the impact of routine standardized CSM on margin status following primary surgery for early stage breast cancer (Stage 0 - II), on post-operative patient satisfaction and cosmetic outcomes, and on general intraoperative time and operative costs. A parallel group format will be implemented to compare this modified surgical therapy - BCS with CSM - with BCS alone, which is the current standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed, biopsy-proven stage 0-II breast cancer.
* Planning to undergo breast-conserving surgery.
* At least 18 years of age and no more than 85 years of age.
* Female.
* Able to understand and willing to sign an IRB-approved written informed consent document.

Exclusion Criteria:

* Prior surgical treatment for this diagnosis.
* Undergone neoadjuvant chemotherapy.
* History of prior chest radiation therapy.
* Known metastatic disease.
* Pregnant.
* Preference for mastectomy instead of breast-conserving surgery.
* History of ipsilateral breast cancer.
* Goggle assessment substudy: Iodine or seafood allergies.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2016-06-13 (Actual); Primary Completion 2019-11-27 (Actual); Study Completion 2019-11-27 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with positive margins on pathological specimen analysis | Completion of surgery for all enrolled patients (approximately 60 months)
Patient perceptions of the surgery as measured by BREAST-Q questionnaire and novel 3-dimensional breast imaging | 6-12 months post-surgery or post-radiation therapy, whichever is later)
  * The BREAST-Q questionnaire consists of 13 sections.
  * The sections ask the patient questions about how they feel about how their breast area looks, how they feel emotionally, any physical side effects, and sexual side effects.
  * Some of the sections ask the patients to answer a question on a scale of None of the Time (equals=1) to All of the Time (equals=5)
  * Some of the sections ask the patients to answer a question on a scale of Very Dissatisfied (equals=1) to Very Satisfied (equals=4)
Compare intraoperative NIR fluorescence from goggle system with pathologic tissue exam results | Completion of surgery for all enrolled patients (approximately 60 months)

SECONDARY OUTCOMES:
Relationship between CSM and volume of tissue excised in association iwth post-operative aesthetic outcomes | 6-12 months post-surgery or post-radiation therapy, whichever is later)
Cost-effectiveness of routine CSM in BCS as measured by operative time, specimen processing, and resource usage | Completion of surgery for all enrolled patients (approximately 60 months)
Disease status associated with cancer biomarkers | Completion of surgery for all enrolled patients (approximately 60 months)
  The investigators plan to assess plasma and serum levels of several candidate biomarkers, including a phosphorylated form of the annexin A2 protein ("P-annexin A2"), in study patients by immunoblotting/ELISA. This biomarker evaluation in the context of disease status will provide new information in the clinical detection and diagnosis of malignancy. Successful validation of these biomarkers may lead to development of novel blood-based cancer diagnostic tests.
Tumor characteristics associated with cancer biomarkers | Completion of surgery for all enrolled patients (approximately 60 months)
  The investigators plan to assess plasma and serum levels of several candidate biomarkers, including a phosphorylated form of the annexin A2 protein ("P-annexin A2"), in study patients by immunoblotting/ELISA. This biomarker evaluation in the context of tumor characteristics will provide new information in the clinical detection and diagnosis of malignancy. Successful validation of these biomarkers may lead to development of novel blood-based cancer diagnostic tests.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Margenthaler, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu